CLINICAL TRIAL: NCT03422549
Title: Diaphragmatic Electrical Activity in Preterm Infants on Non-Invasive High Frequency Oscillatory Ventilation (DEAP-NHFO Study)
Brief Title: Diaphragmatic Electrical Activity in Preterm Infants on Non-Invasive Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jonathan Wong, Neonatologist, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H17-02003
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Respiratory Distress Syndrome, Newborn; Chronic Lung Disease of Newborn (Diagnosis)
Keywords: diaphragm; non-invasive ventilation; high-frequency oscillation; CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Active Comparator): Nasal continuous positive airway pressure is a frequently used modality for non-invasive respiratory support in preterm infants.
  Intervention: Device: Drager VN500 Ventilator
  Interventions: Device: Drager VN500 Ventilator
- NHFOV (Active Comparator): Non-invasive high-frequency ventilation is a relatively new modality that is being utilized to support preterm infants and prevent the need for invasive ventilation, but this particular modality has not been well studied to date.
  Intervention: Device: Drager VN500 Ventilator
  Interventions: Device: Drager VN500 Ventilator

INTERVENTIONS:
Device: Drager VN500 Ventilator — This ventilator is capable of providing both CPAP and NHFOV support.

SUMMARY:
Preterm babies have immature lungs and frequent pauses in their breathing which often necessitates breathing support. Nasal Continuous Positive Airway Pressure (CPAP) is one of the most commonly used tools but does not always provide enough support. A new option is non-invasive high frequency ventilation (NHFOV), which gently shakes the lungs to help with gas exchange and may decrease a baby's work of breathing. The investigators plan to study very low birth weight preterm babies who are generally well but require some support with their breathing. By inserting a special feeding tube with sensors into the stomach, the investigators can measure the electrical activity of the diaphragm (EAdi), which is an important muscle for breathing. By analyzing EAdi in babies receiving either CPAP or NHFOV, the investigators will be able to measure and compare how each method of support affects a baby's breathing. This important study will help us determine the most appropriate breathing support for preterm babies.

DETAILED DESCRIPTION:
Continuous Positive Airway Pressure is one of the most researched and accepted methods of delivering NIV to term and preterm infants. Non-invasive high frequency ventilation is a relatively new method of delivering NIV respiratory support in preterm infants. Preliminary studies suggest superiority over CPAP, and NHFOV is being increasingly utilized in clinical practice in an attempt to prevent intubation and minimize ventilation-induced lung injury in preterm infants. However, little is known about its mechanism of action and its effect on respiratory mechanics in the newborn. The objective of this study is to compare the effects of non-invasive ventilation (NIV) delivered by nasal Continuous Positive Airway Pressure (CPAP) versus Non-Invasive High Frequency Ventilation (NHFOV) on respiratory pattern as assessed by the electrical activity of the diaphragm (EAdi) in very low birth weight (VLBW) preterm infants.

The investigators hypothesize that in VLBW preterm infants with relative pulmonary insufficiency, NHFOV will reduce respiratory drive and improve ventilation, subsequently resulting in decreased patient diaphragm energy expenditure. This would be demonstrated by decreased neural respiratory rates and/or decreased peak electrical activity of the diaphragm while breathing on NHFOV compared to CPAP.

Clinicians are seeking alternative methods for providing non-invasive respiratory support to preterm infants. NHFOV is a relatively new modality that is being increasingly utilized in clinical practice but has not been well studied. This study will help the investigators determine how non-invasive high frequency ventilation affects breathing in preterm infants, as compared to the more traditional modality of nasal CPAP. Therefore, clinicians will not only be able to better understand how NHFOV works, but also utilize this information to decide on the most appropriate respiratory support modality for preterm patients

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable preterm infants with birth weights ≤1500g admitted to the neonatal intensive care unit (NICU) at the Children's and Women's Hospital of BC
* On nasal continuous positive airway pressure of 6 to 8 cmH20 support for at least 48 hours, treated with methylxanthines for apnea of prematurity and requiring 21-40% of oxygen.

Exclusion Criteria:

* infants with congenital anomalies of the gastrointestinal tract, phrenic nerve damage, diaphragmatic paralysis, esophageal perforation.
* infants with congenital or acquired neurological deficit (including significant intraventricular hemorrhage >Grade II), neonatal seizure.
* infants with significant congenital heart disease (including symptomatic PDA).
* infants with congenital anomalies of the diaphragm.
* infants with congenital anomalies of the respiratory tracts (e.g. Congenital Cystic Adenomatoid Malformation (CCAM)).
* infants requiring ongoing treatment for sepsis, necrotizing enterocolitis (NEC), antibiotics for lung infections, narcotic analgesics, or gastric motility agents.
* infants on nasal CPAP and requiring more than 40% oxygen
* infants with significant gastric residuals and vomiting.
* infants with facial anomalies.
* infants with pneumothorax or pneumomediastinum.
* infants in the immediate postoperative period.

Ages: 48 Hours to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the peak electrical activity of the diaphragm between CPAP and NHFOV. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (CPAP and NHFOV).

SECONDARY OUTCOMES:
Difference in neural respiratory rate. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (CPAP and NHFOV).
Difference in neural inspiratory time. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (CPAP and NHFOV).
Difference in diaphragm energy expenditure. | 4 hours
  Measured by the electrical activity of the diaphragm between respiratory support modes (CPAP and NHFOV).
Difference in transcutaneous pCO2 on the different modes of non-invasive ventilation. | 4 hours
  TpCO2 bedside measurement.
Difference in the number of apnea episodes. | 4 hours
  Clinical monitoring and vitals monitoring at the bedside.
Differences in SpO2 histogram classification between modes of ventilation. | 4 hours
  Electronic vitals monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wong, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Women's Hospital and Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided